CLINICAL TRIAL: NCT01069367
Title: Open-label, Uncontrolled Postmarketing Study to Evaluate Immunogenicity, Safety and Tolerability of Cell-derived A/H1N1 Influenza HA Vaccine in Healthy Japanese Elderly Subjects
Brief Title: Open-label, Uncontrolled Postmarketing Study of Cell-derived A/H1N1 Influenza HA Vaccine in Japanese Elderly Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V110_10
Record Dates: First submitted 2010-02-15; First posted 2010-02-17 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2012-01

CONDITIONS: Swine-Origin Influenza A H1N1 Virus
Keywords: Influenza A; H1N1 subtype; Children/adolescent; Vaccine; Adjuvant; Cell culture
MeSH Terms: interventions — Emulsions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm:1 (Experimental)
  Interventions: Biological: Emulsion, Cell Culture-based, influenza HA vaccine H1N1

INTERVENTIONS:
Biological: Emulsion, Cell Culture-based, influenza HA vaccine H1N1 — Cell-derived A/H1N1 influenza HA vaccine (0.25 mL as injection volume)

SUMMARY:
This is to evaluate immunogenicity based on EMEA/CHMP criteria, and safety & tolerability of cell-derived A/H1N1 influenza HA vaccine in healthy Japanese elderly subjects.

DETAILED DESCRIPTION:
This is an open-label, uncontrolled post-marketing study of the cell-derived A/H1N1 influenza HA vaccine. Subjects received 3.75μg of cell-derived H1N1sw vaccine formulated in half (i.e., half the content of the European-licensed adjuvanted seasonal influenza vaccine) MF59 adjuvant (3.75_halfMF59). All vaccination were administered IM in the deltoid muscle, preferably of the non-dominant arm at the first vaccination and of the opposite arm to the first vaccination, as a rule, at the second vaccination. Blood samples were collected at baseline (day1), 3 weeks after the first vaccination (day 22) and three weeks after the second vaccination (day 43). Sera were tested by Hemagglutination Inhibition (HI) assay. Local and systemic reactions were collected for the first week following each injection using Diary Card (i.e. Day 1 to Day 7 and Day 22 to Day 28). All AEs, SAEs, and AEs that led to withdrawal from the study and related prescription medications were collected for the entire study period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese aged over 60 years

Exclusion Criteria:

* Any serious chronic or progressive disease according to judgment of the investigator (including, but not limited to neoplasm, insulin dependent diabetes, cardiac, renal, hepatic or respiratory disease)
* History of any anaphylaxis, serious vaccine reactions, or hypersensitivity to influenza viral proteins, to any excipients
* Administration of swine influenza (A/H1N1) vaccine prior to Day 1 or documented confirmed or suspected swine influenza disease
* History of progressive or sever neurological disorders
* Known or suspected impairment/alteration of immune function

Min Age: 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-03; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Seroprotection, GMRs and Seroconversion rate at Weeks 0, 3 and 6 | 6 weeks

SECONDARY OUTCOMES:
Solicited reactions, AEs, vital signs, laboratory tests | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (1):
- CPC Clinic, Medipolis Medical Research Institute, Kagoshima, Japan

REFERENCES:
- [Result] Fukase H, Furuie H, Yasuda Y, Komatsu R, Matsushita K, Minami T, Suehiro Y, Yotsuyanagi H, Kusadokoro H, Sawata H, Nakura N, Lattanzi M. Assessment of the immunogenicity and safety of varying doses of an MF59(R)-adjuvanted cell culture-derived A/H1N1 pandemic influenza vaccine in Japanese paediatric, adult and elderly subjects. Vaccine. 2012 Jul 13;30(33):5030-7. doi: 10.1016/j.vaccine.2012.03.053. Epub 2012 Apr 1. PMID 22472791